CLINICAL TRIAL: NCT05880953
Title: Parent-to-parent Coaching While Awaiting Hospital Discharge With a Child With a Ventilator: an Empowerment Model for Home Health Nurse (HHN) Advocacy
Brief Title: Parent-to-parent Coaching While Awaiting Hospital Discharge With a Child With a Ventilator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB23-0348; P50MD017349 (NIH)
Record Dates: First submitted 2023-05-11; First posted 2023-05-30 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Invasive Mechanical Ventilation; Children With Medical Complexity; Home Nursing; Empowerment
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent Coaching (Experimental): Participants will be involved for about 6 months or until they feel that they no longer need the parent-to-parent support.
  Parents will participate in the following contact attempts:
  * Introductions and rapport building which will include a demographic survey with a needs assessment, and the Family Empowerment Scale (FES)
  * A series of coaching points which may include some or all of the following topics
    * Interviewing and selecting a home health agency
    * Expectation setting for home based nursing care
    * Tips for finding home health professionals from inpatient nursing
    * Tips for using personal and professional care networks to find and recruit home health team members
  * An exit interview assessment including the FES and components of the demographic survey that may have changed
  Interventions: Behavioral: Parent-to-parent coaching

INTERVENTIONS:
Behavioral: Parent-to-parent coaching — Parents and parent coaches will meet as needed via the family's preferred method. Engagement may include text messaging, phone conferencing, Zoom conferencing, or occasional in-home or hospital visiting as preferred. Coaching sessions will vary based on family desired frequency and location, but may include: on-site in the family home or hospital room, telephone or video conferencing, or asynchronous contacts via email or text messaging. The template for the intervention includes an initial introductory session which is intended to build rapport and orient the parent to our program. Subsequent session topics may include: addressing specific needs including topics of interviewing and selecting home health agencies, expectation setting for home based nursing care, recruiting for home health team from inpatient settings, and recruiting for home health team from professional and personal networks.

SUMMARY:
The objective of the study is to pilot a parent-to-parent coaching model with experienced family members of children with Invasive Mechanical Ventilation (IMV) as parent coaches.

DETAILED DESCRIPTION:
The objective of the study is to pilot a parent-to-parent coaching model with experienced family members of children with IMV as parent coaches. Parent coaches will advise parents of children with IMV awaiting hospital discharge on strategies for advocating for home nursing. Parents and parent coaches will meet as needed and engagement will be tailored to parent preference: text messaging, video or phone conferencing, or in-person visiting in the family home or hospital. Points of contact, issues addressed, and time required will be collected as needs assessment data to appropriately size and scale a future intervention. Enrollment and exit assessments will include completion of the Family Empowerment Scale (FES) and a brief structured interview about parents' perceived impact and acceptability, which will provide pilot data to inform a future intervention. The investigator hypothesizes that parents will gain self-advocacy skills specific to recruiting home health nurses and improve the size of their home nursing workforce through this coaching model.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children with a tracheostomy and ventilator awaiting hospital discharge in Illinois.
* Parents must live or have their child hospitalized within approximately a 1 hour radius of the University of Chicago.
* The child must be enrolled in, or in the process of enrolling in the Division of Specialized Care for Children (DSCC) Home Care Program.
* The parent/legal guardian must have legal custody of the child and plan on living with the child in the home.

Exclusion Criteria:

* Wards of the state

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2025-05-09 (Actual)

PRIMARY OUTCOMES:
Change in parent empowerment as measured by the family empowerment scale (FES) | Baseline and repeated at exit (either at 6 months or when parents choose to exit the study)
  Parents will complete the Family Empowerment Scale (FES), a 34-item scale designed to assess empowerment in parents whose children have emotional disabilities.

SECONDARY OUTCOMES:
Change in nursing coverage | Baseline and repeated at exit (either at 6 months or when parents choose to exit the study)
  Parents will complete REDCap survey indicating their home nursing coverage.
Satisfaction with coaching program | exit (either at 6 months or when parents choose to exit the study)
  Parents will complete a structured interview about their satisfaction with the program.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Sobotka, MD, MSCP, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No Individual Participant Data(IPD) will be shared.